CLINICAL TRIAL: NCT03341949
Title: Soluble CD146 and Proteinuria in Chronic Renal Disease
Acronym: CPinMRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-12; ID RCB (Registry Identifier: 2017-A01046-47)
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with chronic kidney disease (Experimental): Determination of the Cluster of Differentiation 146 (CD146)
  Interventions: Biological: Recurring blood sample

INTERVENTIONS:
Biological: Recurring blood sample — An additional tube will be collected for the assay of CD146s as part of the research

SUMMARY:
Chronic renal disease (CKD) is defined as a decrease in glomerular filtration rate (GFR) and / or proteinuria or albuminuria (a protein present in urine). Albuminuria is considered a marker of endothelial dysfunction. Proteinuria and / or albuminuria are recognized as cardiovascular risk factors in both diabetic and non-diabetic populations, independently of GFR. It is also a marker of progression of kidney disease. cluster of differentiation 146 (CD146) is an endothelial adhesion molecule with preferential localization in the junction. Soluble CD146 (or CD146s). CD146s is a biomarker of endothelial dysfunction that is easy to assay. The increase in CD146 levels was described during the MRC, especially in diabetic patients with significant proteinuria. In two independent cohorts of patients with CDR, CD146s did not correlate with creatinine or GFR but appeared to correlate with proteinuria.

The aim of our study is to determine whether the blood concentration of CD146s is correlated with proteinuria independently of GFR. For this purpose, we propose this study in the kidney nephrology and transplantation center of Conception Hospital, with the objective of highlighting the link between proteinuria and serum CD146 levels in patients with CKD, whatever their renal function and / or underlying pathology. 205 patients will be included over two years with dosing of CD146s and proteinuria at the same time. These 205 patients will be recruited at each stage of the CKD (41 in each arm). CD146s could be a new biomarker predicting the risk of renal function impairment or cardiovascular risk independent of renal function.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject aged 18 years or over
* Subject capable of giving informed consent
* Patient with chronic kidney disease (stage 1 to 5 CKD regardless of etiology)

Exclusion Criteria:

* Pregnant or lactating woman
* Person deprived of liberty or hospitalized without consent
* Major under legal protection or unable to express his consent
* Refusal of the patient
* Patient with a history of kidney transplantation
* Evolutionary cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Serum CD146s assay | 12 months
  determining the blood concentration of CD146s is correlated with proteinuria regardless of glomerular filtration rate (GFR).
The dosage of proteinuria | 12 months
  determining the blood concentration of CD146s is correlated with proteinuria regardless of glomerular filtration rate (GFR).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France